CLINICAL TRIAL: NCT07124364
Title: Comparison of the Effects of Benson Relaxation Technique, Mindfulness-Based Meditation, and Breathing Therapy on Alarm Fatigue and Psychological Well-Being in Intensive Care Nurses: A Four-Arm, Assessor-Blinded, Randomized Controlled Trial
Brief Title: Effects of Relaxation, Mindfulness, and Breathing Therapy on Alarm Fatigue and Psychological Well-being in Intensive Care Nurses
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacer Eroglu (Other)
Collaborators: Ankara City Hospital Bilkent (Other); Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Hacer Eroglu, Assistant Professor, PhD, RN, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Record 5
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Alarm Fatigue in Intensive Care Unit Nurses; Psychological Well-Being in Intensive Care Unit Nurses
Keywords: Alarm fatigue; Psychological well-being; Intensive care nurses; Benson Relaxation Technique; Breathing therapy; Randomized controlled trial; ICU; Nursing intervention
MeSH Terms: conditions — Alert Fatigue, Health Personnel; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Four-arm, assessor-blinded, randomized controlled trial with parallel group assignment.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and the statistician will be blinded to group allocation. Due to the nature of mind-body interventions, participants and intervention providers cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Benson Relaxation Technique Group (Experimental): Participants will receive weekly 30-minute group sessions for 8 weeks to practice the Benson Relaxation Technique under the guidance of a trained instructor. They will also be instructed to perform daily home practice.
  Interventions: Behavioral: Benson Relaxation Technique
- Mindfulness-Based Stress Reduction Meditation Group (Experimental): Participants will attend weekly 30-minute group sessions for 8 weeks, focusing on seated mindfulness meditation and mindful breathing exercises. They will also be encouraged to practice daily at home.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction Meditation
- Breathing Therapy Group (Experimental): Participants will attend weekly 30-minute group sessions for 8 weeks, performing guided breathing exercises designed to reduce stress and promote relaxation. Daily home practice will be encouraged.
  Interventions: Behavioral: Breathing Therapy
- Control Group (No Intervention): Participants will not receive any intervention during the study period and will continue their usual routine. After the study ends, they will be offered the opportunity to participate in one of the intervention programs.

INTERVENTIONS:
Behavioral: Benson Relaxation Technique — The Benson Relaxation Technique is a structured relaxation method involving the repetition of a word, sound, or phrase while sitting quietly in a comfortable position with eyes closed, combined with passive muscle relaxation. In this study, it will be delivered in weekly 30-minute group sessions for 8 weeks by a trained instructor. Participants will be instructed to practice the technique daily at home for 10-15 minutes.
  Arms: Benson Relaxation Technique Group
Behavioral: Mindfulness-Based Stress Reduction Meditation — Mindfulness-Based Stress Reduction meditation is a practice focusing on cultivating awareness of the present moment through seated meditation and mindful breathing. In this study, participants will attend weekly 30-minute group sessions for 8 weeks, guided by an experienced instructor. They will also be encouraged to perform daily mindfulness meditation at home for 10-15 minutes.
  Arms: Mindfulness-Based Stress Reduction Meditation Group
Behavioral: Breathing Therapy — Breathing therapy consists of guided breathing exercises designed to promote relaxation, reduce stress, and improve psychological well-being by regulating breathing patterns. In this study, participants will attend weekly 30-minute group sessions for 8 weeks, led by a trained facilitator. Daily home practice of slow deep breathing techniques for 10-15 minutes will be encouraged.
  Arms: Breathing Therapy Group

SUMMARY:
The goal of this clinical trial is to compare the effects of the Benson Relaxation Technique, mindfulness-based stress reduction meditation, and breathing therapy on reducing alarm fatigue and improving psychological well-being in intensive care unit (ICU) nurses.

The main questions it aims to answer are:

Do the Benson Relaxation Technique, mindfulness-based stress reduction meditation, and breathing therapy significantly reduce alarm fatigue in ICU nurses?

Do these interventions significantly improve psychological well-being in ICU nurses?

Researchers will compare three intervention groups (Benson Relaxation Technique, mindfulness-based stress reduction meditation, breathing therapy) with a control group receiving no intervention to determine which approach produces the greatest improvement in alarm fatigue and psychological well-being.

Participants will:

Attend weekly group sessions for their assigned intervention over the course of [8 weeks].

Practice the assigned technique regularly between sessions as instructed.

Complete questionnaires assessing alarm fatigue and psychological well-being before and after the intervention.

DETAILED DESCRIPTION:
This clinical trial was designed to address a gap in the literature regarding effective mind-body approaches for reducing alarm fatigue and supporting psychological well-being among intensive care unit (ICU) nurses. Alarm fatigue is a common and serious concern in ICUs, and interventions that improve nurses' mental health may also enhance patient safety. In this study, three mind-body-based interventions-Benson Relaxation Technique (BRT), mindfulness-based stress reduction meditation (MBSR), and breathing therapy-will be compared in terms of their effects on alarm fatigue and psychological well-being. The comparative findings from this trial are expected to help identify the most effective mind-body-based approach for ICU nurses and support its wider implementation in clinical practice.

Hypotheses

H₀: BRT, MBSR, and breathing therapy have no significant effect on alarm fatigue and psychological well-being in ICU nurses.

H₁: BRT, MBSR, and breathing therapy have a significant effect on alarm fatigue and psychological well-being in ICU nurses.

Study Design This study will employ a four-arm, assessor-blinded, randomized controlled trial design.

Study Setting and Duration The trial will be conducted at three ICU centers: the Internal Medicine and General Intensive Care Units of Ankara Bilkent City Hospital - General Hospital Tower, and the Internal Medicine ICUs of Hacettepe University Adult and Oncology Hospitals. Data collection will take place between June 2025 and June 2026.

Institutional Characteristics The Internal Medicine and General ICUs of Ankara Bilkent City Hospital - General Hospital Tower are tertiary-level units serving approximately 140-150 patients daily, with a total of 70 ICU nurses. The Internal Medicine ICUs of Hacettepe University Adult and Oncology Hospitals serve approximately 200 patients daily across four units, staffed by a total of 100 ICU nurses.

Population and Sample The study population will consist of nurses working in the above-mentioned tertiary ICUs. The sample will include nurses who meet the inclusion criteria, volunteer to participate, and provide written and verbal informed consent. Sample size was calculated based on a previous randomized controlled trial by Askar et al. (2024) examining the effects of progressive muscle relaxation on fatigue in ICU nurses. In that study, mean fatigue scores at week 4 were 3.13±1.58 for the intervention group and 4.12±1.70 for the control group, with a statistically significant difference between groups. Using these findings, an effect size of 0.62, a 95% confidence level, 88% power, and α = 0.05, the minimum required sample size was determined as 42 nurses per group, totaling 168 participants.

Inclusion Criteria

Age ≥ 18 years

Bachelor's degree or higher in nursing

At least 6 months' experience in a tertiary ICU

Cognitive and physical ability to complete study forms and perform the assigned exercise with the researcher

Voluntary participation with signed informed consent

Exclusion Criteria

Diagnosed psychological disorders requiring treatment (e.g., anxiety, panic disorder, depression)

Not actively working during the study period due to leave (e.g., maternity, annual leave)

Concurrent participation in another relaxation exercise program (e.g., yoga, visualization)

Participants will also be withdrawn if they:

Request to leave the study during the intervention period

Miss two consecutive weekly group sessions

Randomization and Blinding Eligible nurses will be randomly assigned (1:1:1:1) to one of the four study arms using www.randomizer.org by the lead researcher. Allocation results will be shared with the second researcher. Interventions will be delivered by a third researcher, while data collection will be performed by a fourth researcher blinded to group allocation. Data analysis will be conducted by a statistician who is also blinded to allocation. Due to the nature of mind-body interventions, participants and the researcher delivering the interventions cannot be blinded; however, the study will maintain assessor blinding.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Bachelor's degree or higher in nursing
* At least 6 months' experience in a tertiary intensive care unit
* Cognitive and physical ability to complete study forms and perform the assigned exercise with the researcher
* Willingness to participate and provide written informed consent

Exclusion Criteria:

* Diagnosed psychological disorders requiring treatment (e.g., anxiety, panic disorder, depression)
* Not actively working during the study period due to leave (e.g., maternity leave, annual leave)
* Concurrent participation in another relaxation exercise program (e.g., yoga, visualization)
* Withdrawal request during the intervention period
* Missing two consecutive weekly group sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Alarm Fatigue | Baseline, at the end of week 4, at the end of week 8, and at the end of week 10
  Alarm fatigue will be measured using the Turkish version of the Healthcare Technology Foundation's Alarm Fatigue Questionnaire, which assesses frequency and perception of alarm-related fatigue among ICU nurses. Higher scores indicate greater fatigue.
Psychological Well-Being | Baseline, at the end of week 4, at the end of week 8, and at the end of week 10
  Psychological well-being will be assessed using the Turkish version of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS). Higher scores indicate better well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Gok Metin, PhD, RN, Principal Investigator — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Bilkent City Hospital - General Hospital Tower, Internal Medicine and General Intensive Care Units, Ankara, Ankara
  - Hacettepe University Hospital, Ankara, Ankara

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including demographic information, baseline and post-intervention outcome measures) will be shared upon reasonable request to the principal investigator, following publication of the study results. Data will be available for 3 years after publication.
Supporting Information: SAP, ICF
Time Frame: De-identified individual participant data and supporting documents will be available beginning 3 months after publication of the main study results and will remain available for 3 years thereafter.
Access Criteria: Qualified researchers will be able to request access to de-identified participant data, the study protocol, statistical analysis plan, and informed consent form by contacting the principal investigator via email. Requests must include a methodologically sound proposal and a signed data use agreement. Approved researchers will receive the requested data through secure electronic transfer.